CLINICAL TRIAL: NCT04486508
Title: Intermediate-dose Versus Standard Prophylactic Anticoagulation In cRitically-ill pATIents With COVID-19: An opeN Label Randomized Controlled Trial---A Randomized Trial of Atorvastatin vs. Placebo In Critically-ill Patients With COVID-19
Brief Title: Intermediate-dose vs Standard Prophylactic Anticoagulation and Statin vs Placebo in ICU Patients With COVID-19
Acronym: INSPIRATION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Tehran Heart Center (Other); Masih Daneshvari Hospital (Other); Hazrat Rasool Hospital (Other); Modarres Hospital (Other); Firuzgar hospital affiliated to Iran University of Medical Sciences (Other); Imam Khomeini Hospital (Other); Sina Hospital, Iran (Other); Tabriz University of Medical Sciences (Other); Shariati Hospital (Other); Imam Ali Hospital (Unknown); Labbafinejhad Hospital (Other)
Responsible Party: Principal Investigator, Parham Sadeghipour, Associate Professor, Rajaie Cardiovascular Medical and Research Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 99060
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Covid19
Keywords: anticoagulation; statin
MeSH Terms: conditions — COVID-19 | interventions — Heparin; Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: 1:1 multicenter open-label 2x2 factorial design randomized controlled trial with allocation sequence concealment and blinded endpoint adjudication.
Who Masked: Outcomes Assessor
Masking Description: For the first hypothesis, allocation sequence concealment and blinded endpoint adjudication.
  For the second hypothesis, allocation sequence concealment, double-blind medication administration, and blinded endpoint adjudication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intermediate dose anticoagulation (Experimental): Intermediate dose anticoagulation will be the the tested regimen. The anticoagulation regimen will be modified according to weight/ body mass index, and creatinine clearance level (Cl Cr). Enoxaparin will be the primary agent for anticoagulation, with unfractionated heparin reserved only for patients with creatinine clearance of ≤15 mL/min according to Cockcroft-Gault Formula.
  Interventions: Drug: intermediate dose Enoxaparin/ unfractionated heparin
- Standard Prophylaxis (Active Comparator): Standard prophylaxis dose anticoagulation will be the anticoagulation of choice in the control arm. Enoxaparin will be the primary agent for anticoagulation, with unfractionated heparin reserved only for patients with creatinine clearance of ≤15 mL/min according Cockcroft-Gault Formula.
  Interventions: Drug: standard prophylactic dose Enoxaparin/ unfractionated heparin
- Atorvastatin 20 (Experimental): Atorvastatin 20 mg daily will be the statin therapy of choice in the intervention arm
  Interventions: Drug: Atorvastatin 20mg
- Atorvastatin 20 mg Matched placebo (Placebo Comparator): Matching placebo will be used for the control arm
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: intermediate dose Enoxaparin/ unfractionated heparin — Intermediate dose anticoagulation according to creatinine clearance and weight
  Other Names: Intermediate dose anticoagulation
  Arms: Intermediate dose anticoagulation
Drug: standard prophylactic dose Enoxaparin/ unfractionated heparin — Standard prophylaxis anticoagulation according to creatinine clearance and weight
  Other Names: Standard dose prophylaxis anticoagulation
  Arms: Standard Prophylaxis
Drug: Atorvastatin 20mg — Statin
  Other Names: Statin
  Arms: Atorvastatin 20
Drug: Matched placebo — Matched placebo to atorvastatin 20 mg
  Other Names: Statin
  Arms: Atorvastatin 20 mg Matched placebo

SUMMARY:
In a 2x2 factorial design randomized controlled trial, the investigators aim to elaborate the safety and efficacy of two pharmacological regimens on outcomes of critically-ill patients with COVID-19. The first randomization entails open-label assignment to intermediate versus standard dose prophylactic anticoagulation. The investigators hypothesize that intermediate dose compared with standard prophylactic dose anticoagulation will have a superior efficacy with respect to a composite of venous thromboembolism (VTE), requirement for extracorporeal membrane oxygenation (ECMO), or all-cause mortality. The second randomization will be double-blind assignment of the included patients to atorvastatin 20mg daily versus matching placebo. The hypothesis is that statin therapy, compared with placebo, will reduce the composite of VTE, need for ECMO, or all-cause mortality.

DETAILED DESCRIPTION:
Coronavirus disease-2019 (COVID-19) -- a viral illness caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) -- has important manifestations outside the pulmonary parenchyma, including microthrombosis and macrothrombosis, with venous thrombosis being the most common form of thrombotic involvement. Existing studies, depending on the type of outcome assessment and type and dose of prophylaxis, have reported thrombotic events in 7-85% of patients with COVID-19.

However, the optimal antithrombotic regimen in these patients remains uncertain. Although many clinicians continue to consider standard-dose prophylactic anticoagulation, other believe that more intense anticoagulation may reduce the thrombotic events, and improve outcomes. However, limited high-quality data exist to inform clinical practice and the existing guidelines recommendations are mostly based on expert opinion and consensus.

In addition, exuberant inflammatory response is known to play a role in the pathophysiology of acute respiratory distress syndrome (ARDS) and COVID-19. It is possible that the pleiotropic effects of statins, which include anti-inflammatory and antithrombotic effects, prove beneficial in patients with severe COVID-19.

This study plans to investigate the safety and efficacy of two pharmacological regimens on outcomes of critically-ill patients with COVID-19 using a 2x2 factorial design.

First, patients will be assessed for the eligibility criteria for the anticoagulation hypothesis. Those meeting the criteria, will be assigned to intermediate versus standard dose prophylactic anticoagulation. These patients will subsequently be assessed for eligibility for the second randomization, and if meeting the criteria, will be assigned to atorvastatin 20mg/d or matching placebo.

ELIGIBILITY:
Inclusion Criteria for Anticoagulation Hypothesis

1. Adult patients (≥18 years), with polymerase chain reaction (PCR)-confirmed COVID-19 admitted to ICU within 7 days of initial hospitalization , who do not have another firm indication for anticoagulation (such as mechanical valve, high-risk atrial fibrillation (AF), VTE, or left ventricle (LV) thrombus),who are not enrolled in another blinded randomized trial, and are willing to participate in the study and provide informed consent .
2. Estimated survival of at least 24 hours at the discretion of enrolling physician

Exclusion Criteria for Anticoagulation Hypothesis

1. Weight <40 Kilogram (kg)
2. Overt bleeding at the day of enrollment
3. Known major bleeding within 30 days (according to the Bleeding Academic Research Consortium (BARC) definition, Appendix A)
4. Platelet count <50,000/Fl
5. Pregnancy (as confirmed by Beta human chorionic gonadotropin (HCG) testing among female patients <50 years)
6. Patients on Extracorporeal Membrane Oxygenation (ECMO)
7. History of heparin induced thrombocytopenia or immune thrombocytopenia
8. Ischemic stroke within the past 2 weeks
9. Craniotomy/major neurosurgery within the past 3 months
10. Major head or spinal trauma in the past 30 days
11. Known brain metastases or vascular malformations (aneurysm)
12. Presence of an epidural, spinal or pericardial catheter
13. Major surgery other than neurosurgery within 14 days prior to enrollment
14. Coexistence of severe obesity (weight >120 kg or BMI>35 kg/m2 along with severe renal insufficiency defined as creatinine clearance (CrCl) <30 mL/sec)
15. Allergic reaction to study medications
16. Lack or withdrawal of informed consent

Inclusion Criteria for the Statin Randomization

1. Patients enrolled for the anticoagulation randomization
2. Willingness to participation in the study and providing informed consent

Exclusions Criteria for the Statin Randomization

1. Baseline liver function tests> 3 times upper normal limits (ULN) or creatine kinase (CK) >500 U/L
2. Active liver disease (LFT>3 ULN plus histologic finding including cirrhosis or inflammation or necrosis)
3. Routine use of statins prior to the index hospitalization
4. Previous documented statin intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
a composite of acute VTE, arterial thrombosis, treatment with ECMO, or all-cause mortality | 30 days from enrollment
  composite of adjudicated 30-day acute VTE, arterial thrombosis, treatment with extracorporeal membrane oxygenation (ECMO), or all-cause mortality.

SECONDARY OUTCOMES:
Rate of all-cause mortality | 30 days from enrollment
  Patient status regarding to being alive or dead at the end of 30-day follow up
Rate of objectively-confirmed VTE | 30 days from enrollment
  Distal or proximal deep vein thrombosis which has been confirmed by ultrasonography or venography/ PE confirmed by at least one CTPA or lung scan
Ventilator free days | 30 days from enrollment
  Difference between days of ICU stay and days on invasive mechanical ventilation
Rate of major bleeding | 30 days from enrollment
  According to the Bleeding Academic Research Consortium (BARC 3 or 5 bleeding)
Rate of clinically-relevant non-major bleeding | 30 days from enrollment
  Clinically-significant bleeding, not fulfilling criteria for major bleeding)
Rate of severe thrombocytopenia | 30 days from enrollment
  Platelet count <20.000
Rate of rise in liver enzymes | 30 days from enrollment
  Increase liver function tests 3 times greater than upper limit of normal
Clinically-diagnosed myopathy | 30 days from enrollment
  Assessed by clinical and biomarker tests according to the treating physicians.
Objectively-confirmed arterial thrombosis | 30 days from enrollment
  Imaging confirmed acute arterial thrombosis (by ultrasonography, CT, MRI, or invasive angiography)

OTHER OUTCOMES:
Rate of objectively clinically-diagnosed type I acute myocardial infarction | 30 days from enrollment
  According to the fourth universal definition of myocardial infraction and confirmed by coronary angiography, intravascular imaging or autopsy
Rate of objectively clinically -diagnosed stroke | 30 days from enrollment
  Any stroke episode which has been confirmed with appropriate diagnostic imaging (brain CT and/or brain MRI)
Rate of objectively clinically -diagnosed acute peripheral arterial thrombosis | 30 days from enrollment
  Imaging confirmed acute peripheral arterial thrombosis (by ultrasonography, CT, MRI, or invasive angiography)
Median ICU length of stay | 30 days from enrollment
  Number of days that a patient has stayed in the ICU
ICU discharge status | 30 days from enrollment
  Status of patients regarding to mortality (alive/dead) at the time of discharge from ICU
Incident atrial fibrillation | 30 days from enrollment
  Any AF episode which has been confirmed by at least one ECG or telemetry monitoring, in patients without prior history of AF
Rate of need for renal replacement therapy | 30 days from enrollment
  Use hemodialysis or veno-venous hemofiltration or peritoneal dialysis for a patient during the hospitalization period, due to acute kidney injury
Post-COVID-19 Functional Status | 60 and 90 -day
  Based on Post-COVID-19 Functional Status questionnaire, which varies fro score 0 to 4, and higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Parham Sadeghipour, MD, Principal Investigator — Rajaie Cardiovascular Medical and Research Center; Behnood Bikdeli, MD, MS, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Masih Daneshvari Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bikdeli B, Talasaz AH, Rashidi F, Sharif-Kashani B, Farrokhpour M, Bakhshandeh H, Sezavar H, Dabbagh A, Beigmohammadi MT, Payandemehr P, Yadollahzadeh M, Riahi T, Khalili H, Jamalkhani S, Rezaeifar P, Abedini A, Lookzadeh S, Shahmirzaei S, Tahamtan O, Matin S, Amin A, Parhizgar SE, Jimenez D, Gupta A, Madhavan MV, Parikh SA, Monreal M, Hadavand N, Hajighasemi A, Maleki M, Sadeghian S, Mohebbi B, Piazza G, Kirtane AJ, Lip GYH, Krumholz HM, Goldhaber SZ, Sadeghipour P. Intermediate versus standard-dose prophylactic anticoagulation and statin therapy versus placebo in critically-ill patients with COVID-19: Rationale and design of the INSPIRATION/INSPIRATION-S studies. Thromb Res. 2020 Dec;196:382-394. doi: 10.1016/j.thromres.2020.09.027. Epub 2020 Sep 24. PMID 32992075
- [Derived] Talasaz AH, Sadeghipour P, Bakhshandeh H, Sharif-Kashani B, Rashidi F, Beigmohammadi MT, Moghadam KG, Rezaian S, Dabbagh A, Sezavar SH, Farrokhpour M, Abedini A, Aliannejad R, Riahi T, Yadollahzadeh M, Lookzadeh S, Rezaeifar P, Matin S, Tahamtan O, Mohammadi K, Zoghi E, Rahmani H, Hosseini SH, Mousavian SM, Abri H, Sadeghipour P, Baghizadeh E, Rafiee F, Jamalkhani S, Amin A, Mohebbi B, Parhizgar SE, Soleimanzadeh M, Aghakouchakzadeh M, Eslami V, Payandemehr P, Khalili H, Talakoob H, Tojari T, Shafaghi S, Tabrizi S, Kakavand H, Kashefizadeh A, Najafi A, Jimenez D, Gupta A, Madhavan MV, Sethi SS, Parikh SA, Monreal M, Hadavand N, Hajighasemi A, Ansarin K, Maleki M, Sadeghian S, Barco S, Siegerink B, Spatz ES, Piazza G, Kirtane AJ, Tassell BWV, Lip GYH, Klok FA, Goldhaber SZ, Stone GW, Krumholz HM, Bikdeli B. Atorvastatin versus Placebo in ICU Patients with COVID-19: Ninety-day Results of the INSPIRATION-S Trial. Thromb Haemost. 2023 Jul;123(7):723-733. doi: 10.1055/a-2059-4844. Epub 2023 Mar 21. PMID 36944357
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Erdem S, Ipek F, Bars A, Genc V, Erpek E, Mohammadi S, Altinata A, Akar S. Investigating the effect of macro-scale estimators on worldwide COVID-19 occurrence and mortality through regression analysis using online country-based data sources. BMJ Open. 2022 Feb 14;12(2):e055562. doi: 10.1136/bmjopen-2021-055562. PMID 35165110
- [Derived] INSPIRATION-S Investigators. Atorvastatin versus placebo in patients with covid-19 in intensive care: randomized controlled trial. BMJ. 2022 Jan 7;376:e068407. doi: 10.1136/bmj-2021-068407. PMID 34996756
- [Derived] INSPIRATION Investigators; Sadeghipour P, Talasaz AH, Rashidi F, Sharif-Kashani B, Beigmohammadi MT, Farrokhpour M, Sezavar SH, Payandemehr P, Dabbagh A, Moghadam KG, Jamalkhani S, Khalili H, Yadollahzadeh M, Riahi T, Rezaeifar P, Tahamtan O, Matin S, Abedini A, Lookzadeh S, Rahmani H, Zoghi E, Mohammadi K, Sadeghipour P, Abri H, Tabrizi S, Mousavian SM, Shahmirzaei S, Bakhshandeh H, Amin A, Rafiee F, Baghizadeh E, Mohebbi B, Parhizgar SE, Aliannejad R, Eslami V, Kashefizadeh A, Kakavand H, Hosseini SH, Shafaghi S, Ghazi SF, Najafi A, Jimenez D, Gupta A, Madhavan MV, Sethi SS, Parikh SA, Monreal M, Hadavand N, Hajighasemi A, Maleki M, Sadeghian S, Piazza G, Kirtane AJ, Van Tassell BW, Dobesh PP, Stone GW, Lip GYH, Krumholz HM, Goldhaber SZ, Bikdeli B. Effect of Intermediate-Dose vs Standard-Dose Prophylactic Anticoagulation on Thrombotic Events, Extracorporeal Membrane Oxygenation Treatment, or Mortality Among Patients With COVID-19 Admitted to the Intensive Care Unit: The INSPIRATION Randomized Clinical Trial. JAMA. 2021 Apr 27;325(16):1620-1630. doi: 10.1001/jama.2021.4152. PMID 33734299
- See also: COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review — https://pubmed.ncbi.nlm.nih.gov/32311448/
- See also: Pharmacological Agents Targeting Thromboinflammation in COVID-19: Review and Implications for Future Research — https://pubmed.ncbi.nlm.nih.gov/32473596/